CLINICAL TRIAL: NCT03192930
Title: Inflammatoriska Och Neurokemiska förändringar Vid ökat Omgivningstryck
Brief Title: Inflammatory and Cerebrospinal Biochemical Markers in Blood During Prolonged Hyperbaric Exposure
Acronym: Mättnad2017
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Swedish Armed Forces Diving and Naval Medicine Centre (Other); KTH Royal Institute of Technology (Other)
Responsible Party: Principal Investigator, Anders Rosén, MD PhD student, Sahlgrenska University Hospital
Other Study IDs: EPN 022-17
Record Dates: First submitted 2017-06-14; First posted 2017-06-20 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2018-03

CONDITIONS: Saturation Exposure; Decompression Injury
Keywords: Hyperbaric; Saturation; Decompression injury; Decompression sickness; Inflammation; Central nervous system injury; Diving medicine
MeSH Terms: conditions — Decompression Sickness; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum. Plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Saturation: Individuals exposed to prolonged hyperbaric exposure
  Interventions: Other: Hyperbaric exposure
- Control: Individuals not exposed to prolonged hyperbaric exposure

INTERVENTIONS:
Other: Hyperbaric exposure — Hyperbaric exposure 4 ATA for 36 hours followed by 70 hours decompression
  Groups: Saturation

SUMMARY:
Research hypothesis

* Prolonged hyperbaric exposure will affect the central nervous system
* Prolonged hyperbaric exposure will induce inflammatory changes
* Prolonged hyperbaric exposure will affect fluid regulation in the body

Objectives:

* To investigate the presence of cerebrospinal biochemical markers in blood during prolonged hyperbaric exposure
* To investigate changes in the quantity of cerebrospinal biochemical markers in blood during decompression after prolonged hyperbaric exposure
* To investigate the presence of inflammatory markers in blood during prolonged hyperbaric exposure
* To investigate changes in the quantity of inflammatory markers in blood during decompression after prolonged hyperbaric exposure
* To investigate if prolonged hyperbaric exposure alters fluid balance in the body

DETAILED DESCRIPTION:
When diving with compressed air, a continuous accumulation of nitrogen will take place in the body. The total uptake of nitrogen by the tissues is dependent on the duration and depth of the performed dive. During prolonged exposure to hyperbaric conditions the body eventually will become saturated with nitrogen. In a hyperbaric environment corresponding to a depth of 30 meters seawater, nitrogen saturation could be expected after about 24 hours. Decompression can cause accumulated nitrogen to form intravascular bubbles.

It has long been considered that decompression sickness (DCS) is caused by bubble formation when dissolved nitrogen at the end of diving comes out of solution. Doppler ultrasound techniques have shown that intravascular gas bubbles could exist even after uneventful dives. Therefore, additional pathophysiological factors must be sought.

Dehydration is a common finding after diving in water. It is probably caused by a combination of a non-existent water intake during diving and a physiologically increased urine production, caused by the increased ambient pressure.

There is evidence of an increased inflammatory activity in blood after diving. Signs of neutrophil activation is a common finding. It is not known if hyperbaric exposure in itself is enough to elicit these biochemical changes or if the presence of intravascular nitrogen bubbles is needed.

Studies have shown that biochemical markers of central nervous system (CNS) injury can be detected in blood samples obtained from patients with DCS, metabolic and neurologic disease, during cardiac surgery and after traumatic brain injuries. Such markers can also be seen in blood after sport activities like boxing and breath hold diving. If biochemical markers of CNS injury will be present in blood after hyperbaric exposure is not known.

Diving is a common activity in society. It is practised both recreationally and professionally. The police, coast guard, emergency services and armed forces employ professional divers.

The Swedish armed forces (SwAF) Diving and Naval Medicine Center (DNC) is responsible for education and training of divers for SwAF. The centre is also responsible for research and development and conduct tests for diving medicine, and tests of underwater equipment.

SwAF DNC will during 2017 perform saturation diving tests in a dry chamber environment. The study "Inflammatory and cerebrospinal biochemical markers in blood during prolonged hyperbaric exposure - an observational controlled study" will be followed out during these tests. It entails venous blood sampling, spirometric testing and cardiac ultrasound.

This is a prospective, controlled observational study. The study aims to involve at least 16 study subjects. Half of the subjects (at least 8 persons), named the intervention group, will be exposed to hyperbaric conditions. The hyperbaric exposure is part of the Swedish navy saturation diving tests. Half of the subjects (at least 8 persons), named the control group, will experience no hyperbaric exposure.

The intervention group will be compressed in a dry hyperbaric chamber to 4 ATA and remain at that pressure for 36 hours. They will then be decompressed 0,5 meters/hour for 30 hours, after which they will be decompressed 0,375 meters/hour for 40 hours. After 70 hours of decompression normal atmospheric pressure will be reached and the subjects will leave the hyperbaric chamber. The oxygen partial pressure inside the chamber will be actively controlled and never exceed 50 kPa.

Members of the intervention group will be examined by a physician trained in diving medicine before and after the hyperbaric exposure. Spirometric testing of lung function will be carried out at both these occasions. Immmediately after hyperbaric exposure cardiac ultrasound will be used to assess presence and duration of VGE.

Five blood samples (6 mL blood each) will be obtained from all study subjects from both groups according to the following plan:

* before compression commences
* about one hour before decompression commences
* within one hour after leaving the hyperbaric chamber
* about 24 hours after leaving the hyperbaric chamber
* if possible, about 5-7 days after leaving the hyperbaric chamber.

Blood samples are obtained from the control group at the same time points as from the intervention group.

In addition to above mentioned samples, blood samples (6 mL blood each) regarding fluid balance will be obtained from intervention group subjects before, during and after hyperbaric exposure.

Signs of DCS will be actively sought.

ELIGIBILITY:
Inclusion Criteria:

* Submariners and divers employed by the Swedish navy or individuals approved by the Swedish navy for work in a hyperbaric Environment.
* Subjects in the intervention group must be participating in the Swedish navy saturation diving tests.

Exclusion Criteria:

- As this is a highly selected population there is no exclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Submariners and divers employed by the Swedish navy and individuals approved by the Swedish navy for work in a hyperbaric environment participating in the Swedish navy saturation diving tests.
  Submariners and divers employed by the Swedish navy and individuals approved by the Swedish navy for work in a hyperbaric environment not participating in the Swedish navy saturation diving tests.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Concentration of inflammatory and cerebrospinal biochemical markers in blood | 14 days
  E. g: tau, NfL, GFAP, UCHL-1, VCAM-1, ICAM-1, Endothemin-1 and others

SECONDARY OUTCOMES:
Biochemical signs of altered fluid balance in the body | 7 days
  Hematocrit
Changes in lung function | 7 days
  Spirometry (FVC, FEV, diffusing capacity)
Presence of Venous gas Emboli (VGE) | 7 days
  Doppler and 2-D echocardiography
Decompression sickness (DCS) | 7 days
  Clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Zetterberg, PhD, Study Director — Göteborg University
Locations (1):
- Gothenburg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosen A, Gennser M, Oscarsson N, Kvarnstrom A, Sandstrom G, Blennow K, Seeman-Lodding H, Zetterberg H. Biomarkers of neuronal damage in saturation diving-a controlled observational study. Eur J Appl Physiol. 2020 Dec;120(12):2773-2784. doi: 10.1007/s00421-020-04499-y. Epub 2020 Sep 25. PMID 32975632